CLINICAL TRIAL: NCT01636661
Title: Safety of Transcranial Direct Current Stimulation in Pediatric Hemiparesis
Acronym: tDCS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Minnesota Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1205M13901
Record Dates: First submitted 2012-06-11; First posted 2012-07-10 (Estimated); Results first posted 2015-07-20 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-10

CONDITIONS: Hemiparesis
MeSH Terms: conditions — Paresis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcranial Direct Current Stimulation (Experimental): Receiving active tDCS
  Interventions: Device: tDCS
- Sham tDCS (Sham Comparator): tDCS equipment set to placebo setting.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — transcranial direct current stimulation- non-invasive brain stimulation
  Other Names: transcranial direct current stimulation

SUMMARY:
The primary objective of this proposal is to investigate the safety of use of transcranial Direct Current Stimulation (tDCS)in children with hemiparesis.

The research question, "Is transcranial Direct Current Stimulation safe for use in children with congenital hemiparesis?" relates to two hypotheses:

1. tDCS will not produce a major adverse event, including seizure activity.
2. No change in paretic or nonparetic hand function or cognitive status will occur.

DETAILED DESCRIPTION:
Completing a pilot safety study is paramount to the future goal of incorporating the tDCS pediatric safety data and combining tDCS and rehabilitation with constraint-induced movement therapy in order to improve motor outcomes beyond what rehabilitation therapies alone can provide and enhance quality of life for these children with hemiparesis.

ELIGIBILITY:
Inclusion Criteria:

1. Congenital Hemiparesis confirmed by most recent MRI or CT radiologic report.
2. Hemispheric Stroke or Periventricular Leukomalacia
3. Ages 8-17 years old
4. ≥ 10 degrees of active motion at the metacarpophalangeal joint
5. Adequate receptive language function to follow two-step commands as evidenced by performance on TOKEN test of intelligence
6. No evidence of seizure activity within the last 2 years.
7. Subject is able to give informed assent and providing a signature, along with the informed consent signature of the legal guardian as evidenced by signature.

Exclusion Criteria:

1. Metabolic Disorders
2. Neoplasm
3. Epilepsy
4. Disorders of Cellular Migration and Proliferation
5. Acquired Traumatic Brain Injury
6. Expressive Aphasia
7. Pregnancy
8. Indwelling metal or incompatible medical devices
9. Evidence of skin disease or skin abnormalities
10. Botulinum toxin or phenol intramuscular block within the one-month preceding tDCS

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2012-07; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette Gillick, PhD, MS, PT, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Gillick BT, Feyma T, Menk J, Usset M, Vaith A, Wood TJ, Worthington R, Krach LE. Safety and feasibility of transcranial direct current stimulation in pediatric hemiparesis: randomized controlled preliminary study. Phys Ther. 2015 Mar;95(3):337-49. doi: 10.2522/ptj.20130565. Epub 2014 Nov 20. PMID 25413621

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: If a child did not exhibit a motor evoked potential from the ipsilesional cortex, they were excluded from the trial after enrollment but before assignment to a group.
Period: Overall Study
Arm/Group | Transcranial Direct Current Stimulation | Sham tDCS
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Pilot study estimating a sample of children with hemiparesis. No formal sample size nor power analysis was performed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Transcranial Direct Current Stimulation | Sham tDCS | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 6 | 11
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 10.7 (3.2) | 16.9 (2.6) | 14.7 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events/Safety Assessment.
Description: Assessment of safety of use of tDCS in children with hemiparesis through vital signs, physician evaluation, subject report of symptoms. Reported are the number of participants who met the following criteria:
  1. Vital Signs (either resting blood pressure or heart rate)- Any greater than 2SD of change in vital signs from pretest to posttest.
  2. Physician Evaluation- Child identified as declining in function from pretest to posttest.
  3. Subject Report of Symptoms- Reports of serious adverse event/symptoms from pretest to posttest.
  Detailed adverse events are reported in the adverse events module.
Time Frame: Baseline, Posttest, Follow-Up Session at One-Week
Population: Pilot study therefore no sample size analysis. Completed per protocol.
Measure: Number; unit: Participants
Arm/Group | Transcranial Direct Current Stimulation | Sham tDCS
Number analyzed (Participants) | 5 | 6
Participants
  Any Change in Vital Signs | 0 | 0
  Decline in Physician Evaluation | 0 | 0
  Reported Serious Adverse Events | 0 | 0

2. Secondary Outcome: Hand Function Decline as Measured by Number of Participants
Description: Measured by the Box and Blocks Test and Grip Strength
Time Frame: Baseline, Posttest, Follow-Up Session at One-Week
Measure: Number; unit: participants
Arm/Group | Transcranial Direct Current Stimulation | Sham tDCS
Number analyzed (Participants) | 5 | 6
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Transcranial Direct Current Stimulation | Sham tDCS
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 1/5 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcranial Direct Current Stimulation (N=5) | Sham tDCS (N=6)
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Reports of tingling under the electrodes. Assessed verbally by participant feedback at scheduled intervals: pre/post and follow-up sessions.
Burning (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sleepiness (Nervous system disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No